CLINICAL TRIAL: NCT00264498
Title: A Randomized, Open-Label Phase II Study Of ZD1839 (IRESSA™) Versus Gemcitabine And Carboplatin In Chemotherapy-Naive Patients With Advanced (Stage IIIB OR IV) Non-Small Cell Lung Cancer And ECOG Performance Status 2
Brief Title: Phase II Iressa & Carbo/Gem in NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0551
Record Dates: First submitted 2005-12-12; First posted 2005-12-13 (Estimated); Results first posted 2009-08-03 (Estimated); Last update posted 2009-08-03 (Estimated); Status verified 2009-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-Small-Cell Lung Cancer; NSCLC; Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Gefitinib; Gemcitabine; Carboplatin

ARMS (2):
- 1 (Active Comparator): Gemcitabine + Carboplatin
  Interventions: Drug: Gemcitabine; Drug: Carboplatin
- 2 (Experimental): Gefitinib
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — oral tablet
  Other Names: IRESSA; ZD1839
  Arms: 2
Drug: Gemcitabine — intravenous injection
  Other Names: Gemzar
  Arms: 1
Drug: Carboplatin — intravenous injection
  Other Names: CBDCA
  Arms: 1

SUMMARY:
The primary objective is to demonstrate in chemotherapy naïve patients with advanced (Stage IIIB or IV) NSCLC and ECOG PS 2 non-inferiority in progression free survival (PFS) for ZD1839 compared to gemcitabine/carboplatin.

ELIGIBILITY:
Inclusion Criteria:

* Advanced Non Small cell Lung Cell Lung cancer
* Never received chemotherapy
* Up and about 50% of waking hours

Exclusion Criteria:

* Spread of lung cancer to the brain
* Low level of white blood cells
* Radiotherapy within 4 weeks

Patients were entered to this study, initiated in 2004, before the significance of predictive factors such as smoking history, adenocarcinoma histology and mutation status was described.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2004-10; Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Canada Oncology Medical Director, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 2 Canadian cancer clinics between October 2004 and October 2007.
Pre-assignment Details: Following enrolment there was a 7 - 28 day screening period, after which if all inclusion/exclusion criteria were met, patients were randomized to treatment.
  Following objective disease progression on randomized treatment (Period 1), subjects were encouraged to crossover to the other treatment (Period 2).
Groups:
- Active Comparator: Gemcitabine + Carboplatin
- Experimental: Gefitinib
Period: Randomized Treatment
Arm/Group | Active Comparator | Experimental
Started | 17 | 18
Completed | 0 (Treatment is not for a fixed period and continues until a discontinuation criterion is met.) | 0 (Treatment is not for a fixed period and continues until a discontinuation criterion is met.)
Not Completed | 17 | 18
Not completed — Death | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Objective disease Progression | 13 | 14
Not completed — Physician Decision | 1 | 0
Not completed — Incorrectly randomized | 1 | 0
Not completed — Study Closure | 1 | 0
Not completed — Protocol Violation | 1 | 0
Period: Crossover Treatment
Arm/Group | Active Comparator | Experimental
Started | 6 | 9
Completed | 0 (Treatment is not for a fixed period and continues until a discontinuation criterion is met.) | 0 (Treatment is not for a fixed period and continues until a discontinuation criterion is met.)
Not Completed | 6 | 9
Not completed — Death | 1 | 3
Not completed — Objective disease progression | 4 | 5
Not completed — Study closure | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator | Experimental | Total
Number analyzed (Participants) | 17 | 18 | 35
Age Continuous [Mean (Standard Deviation); unit: Years]
  Age at screening | 67.8 (6.01) | 66.2 (8.24) | 67.0 (7.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8.0 | 6.0 | 14.0
  Male | 9.0 | 12.0 | 21.0
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 16.0 | 12.0 | 28.0
  Black | 1.0 | 0 | 1.0
  Oriental | 0 | 4.0 | 4.0
  Other | 0.0 | 2.0 | 2.0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Interval between date of randomization and earliest date of objective disease progression per RECIST criteria or death due to any cause in the absence of progression
Time Frame: Date of randomization to earliest date of objective disease progression
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Active Comparator | Experimental
Number analyzed (Participants) | 17 | 18
Days | 131.0 (66.0000) [66.0 to 190.0] | 42.0 (35.0000) [35.0 to 90.0]

ADVERSE EVENTS:
Arm/Group | Active Comparator | Experimental
Serious Adverse Events (participants affected / at risk) | 4 | 4
Other Adverse Events (participants affected / at risk) | 23 | 26
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Active Comparator | Experimental
Febrile Neutropenia (Blood and lymphatic system disorders) | 1/23 | 0/26
Cardio-Respiratory Arrest (Cardiac disorders) | 0/23 | 1/26
Vomiting (Gastrointestinal disorders) | 1/23 | 0/26
Pneumonia (Infections and infestations) | 1/23 | 2/26
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0/23 | 1/26
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1/23 | 0/26
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1/23 | 0/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Active Comparator | Experimental
Neutropenia (Blood and lymphatic system disorders) | 7/23 | 0/26
Anaemia (Blood and lymphatic system disorders) | 2/23 | 0/26
Thrombocytopenia (Blood and lymphatic system disorders) | 2/23 | 0/26
Diarrhoea (Gastrointestinal disorders) | 2/23 | 14/26
Nausea (Gastrointestinal disorders) | 11/23 | 8/26
Vomiting (Gastrointestinal disorders) | 1/23 | 7/26
Constipation (Gastrointestinal disorders) | 12/23 | 3/26
Stomatitis (Gastrointestinal disorders) | 2/23 | 3/26
Dyspepsia (Gastrointestinal disorders) | 2/23 | 2/26
Abdominal pain (Gastrointestinal disorders) | 1/23 | 2/26
Abdominal distension (Gastrointestinal disorders) | 2/23 | 0/26
Toothache (Gastrointestinal disorders) | 2/23 | 0/26
Fatigue (Gastrointestinal disorders) | 10/23 | 6/26
Asthenia (Gastrointestinal disorders) | 5/23 | 6/26
Oedema peripheral (Gastrointestinal disorders) | 3/23 | 3/26
Pyrexia (Gastrointestinal disorders) | 1/23 | 3/26
Chest pain (Gastrointestinal disorders) | 0/23 | 3/26
Catheter site pain (Gastrointestinal disorders) | 3/23 | 1/26
Pain (Gastrointestinal disorders) | 3/23 | 0/26
Pitting oedema (Gastrointestinal disorders) | 2/23 | 0/26
Urinary tract infection (Infections and infestations) | 0/23 | 2/26
Upper respiratory tract infection (Infections and infestations) | 2/23 | 1/26
Weight decreased (Infections and infestations) | 2/23 | 2/26
Anorexia (Metabolism and nutrition disorders) | 2/23 | 4/26
Decreased appetite (Metabolism and nutrition disorders) | 0/23 | 4/26
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4/23 | 2/26
Back pain (Musculoskeletal and connective tissue disorders) | 2/23 | 2/26
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0/23 | 2/26
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2/23 | 1/26
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2/23 | 1/26
Headache (Nervous system disorders) | 5/23 | 4/26
Hypoaesthesia (Nervous system disorders) | 0/23 | 4/26
Dizziness (Nervous system disorders) | 4/23 | 2/26
Somnolence (Nervous system disorders) | 2/23 | 0/26
Insomnia (Psychiatric disorders) | 1/23 | 3/26
Anxiety (Psychiatric disorders) | 2/23 | 2/26
Confusional state (Psychiatric disorders) | 2/23 | 2/26
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10/23 | 9/26
Cough (Respiratory, thoracic and mediastinal disorders) | 4/23 | 6/26
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2/23 | 3/26
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 3/23 | 2/26
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2/23 | 2/26
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0/23 | 2/26
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6/23 | 1/26
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3/23 | 1/26
Rash (Skin and subcutaneous tissue disorders) | 3/23 | 6/26
Pruritus (Skin and subcutaneous tissue disorders) | 1/23 | 5/26
Dry skin (Skin and subcutaneous tissue disorders) | 0/23 | 4/26
Erythema (Skin and subcutaneous tissue disorders) | 2/23 | 2/26
Acne (Skin and subcutaneous tissue disorders) | 0/23 | 2/26
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2/23 | 1/26
Alopecia (Skin and subcutaneous tissue disorders) | 2/23 | 0/26

LIMITATIONS AND CAVEATS:
No analysis of the efficacy results was performed as the study was prematurely terminated with only 35 out of the planned 122 subjects randomized.

Serious and Other adverse event data for Periods 1 and 2 were combined by treatment for this report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days